CLINICAL TRIAL: NCT00345410
Title: A Randomized, Double-Blind, Parallel-Group, Placebo-Controlled, Multicenter Study Evaluating the Efficacy and Safety of Three Doses of AVE1625 in Abdominally Obese Patients With Atherogenic Dyslipidemia
Brief Title: Dose-Ranging Study Evaluating AVE1625 in Abdominally Obese Patients With Atherogenic Dyslipidemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DRI6412
Record Dates: First submitted 2006-06-27; First posted 2006-06-28 (Estimated); Last update posted 2008-12-19 (Estimated); Status verified 2008-12

CONDITIONS: Obesity; Dyslipidemia
Keywords: obesity and dyslipidemia
MeSH Terms: conditions — Obesity; Dyslipidemias

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: AVE1625 B

SUMMARY:
Primary objective: to assess the effect of AVE1625 on weight loss over a period of 24 weeks in abdominally obese patients with atherogenic dyslipidemia. Secondary objectives: - To assess the dose effect relationship of AVE1625 on HDL-cholesterol and triglycerides plasma levels over a period of 24 weeks - To assess the efficacy of AVE1625 on secondary parameters such as waist circumference and other metabolic parameters over a period of 24 weeks - To assess the safety and tolerabillity of AVE1625 over a period of 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Abdominal obese patients with ·
* Waist circumference > 102 cm in men and >88 cm in women
* Dyslipidemia consisting of :

  * Triglycerides ≥ 1.50 g/L (i.e 1.69 mmol/L) and ≤ 7.0 g/L(i.e. 7.90 mmol/L)AND/OR
  * HDL-cholesterol < 50 mg/dL (i.e. 1.29 mmol/L) in women and < 40 mg/dL (i.e. 1.04 mmol/L) in men

Exclusion Criteria:

* Pregnancy or lactation
* Women of child-bearing potential with no medically approved contraception
* Patients with type 1 diabetes
* Patients with type 2 diabetes must be on a stable dose of oral antidiabetic drugs (excluding glitazones, exenatide, sulfonylurea and nateglinide) and should not receive insulin therapy
* Patients with any clinically significant endocrine disease
* Patients on anticoagulants (heparin, warfarin) or with bleeding disorders
* Clinically relevant disease interfering with subject's safety or making implementation of the study protocol or interpretation of study results difficult
* Patients with mental retardation or any clinically significant psychiatric disorder
* History or concurrent substance abuse (other than nicotine or caffeine especially marijuana or hashish)
* Chronic systemic corticotherapy
* Patients with weight change > 5kg within 3 months prior to screening
* Patients should not have received anti-obesity drugs or other drugs for weight reduction in the 3 months prior to screening.
* The investigator will evaluate whether there are other reasons why a patient may not participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 345 (Actual)
Dates: Start 2006-06; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Absolute change from baseline in body weight at 24 weeks

SECONDARY OUTCOMES:
- relative change from baseline to 24 weeks in plasma HDL-cholesterol and triglycerides levels ; - change from baseline to 24 weeks in waist circumference ; Other criteria: glycemic control parameters.
Safety: physical examination, vital signs, adverse events, ECG, laboratory tests.
Pharmacokinetics: plasma AVE1625 concentrations

CONTACTS AND LOCATIONS:
Overall Officials: Julio ROSENSTOCK, MD, Principal Investigator — Dallas Diabetes and Endocrine Center 7777 Forest Lane, C-618 Dallas TX 75230 USA
Locations (1):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States

REFERENCES:
- See also: Related Info — http://www.sanofi-aventis.com